CLINICAL TRIAL: NCT02386735
Title: Reduction of Corticosteroid Use in Outpatient Treatment of Exacerbated COPD - a Randomized, Double-blind, Non-inferiority Study (The "RECUT"-Trial)
Brief Title: Reduction of Corticosteroid Use in Outpatient Treatment of Exacerbated COPD
Acronym: RECUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate, motivation and engagement of participating GPs unfortunately declined over time, as well as the financial resources.
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Collaborators: Institut für Hausarztmedizin Basel (Unknown); Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Prof. Dr. med., Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSBL2015-017
Record Dates: First submitted 2015-02-11; First posted 2015-03-12 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Adverse Effect of Glucocorticoids and Synthetic Analogues; Disease Exacerbation
Keywords: Corticosteroid treatment; COPD; Primary Health Care; Randomized controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational treatment (Experimental): Patients included in the placebo group are receiving systemic corticosteroid treatment (equivalent of 40mg prednisone daily) for three days followed by two days of placebo.
  Interventions: Drug: Placebo
- Standard treatment (Active Comparator): Patients included in the control group are receiving systemic corticosteroid treatment (equivalent of 40mg prednisone daily) for five days as recommended in current guidelines.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Placebo — Three days prednisone 40mg, two days placebo
  Arms: Investigational treatment
Drug: Prednisone — Five days prednisone 40mg.
  Arms: Standard treatment

SUMMARY:
Background

Chronic obstructive pulmonary disease (COPD) is a major public health issue with no curative treatment. In Switzerland estimated 5-7% of the total population are suffering from this chronic disease. According to current guidelines corticosteroids are part of treatment of acute exacerbations in COPD patients. Several studies suggest that corticosteroids accelerate the recovery of forced expiratory volume in 1 second (FEV1), decrease duration of hospitalization, reduce treatment failure rate and improve clinical outcome. The additional therapeutic benefit on FEV1-recovery tough seems only to last for three to five days. The investigators recently published a hospital-based study showing that in patients presenting to emergency departments with acute exacerbation of COPD, a short five day treatment with systemic steroids was not inferior to a conventional 14 day treatment with regard to re-exacerbation. Cumulative corticosteroid dose could be reduced in this trial. To the investigators knowledge no data is available about the minimal necessary corticosteroid dose in an outpatient treatment setting so far.

Aim

The primary aim of this study is to investigate in an outpatient setting, whether a three day treatment with orally administered systemic corticosteroids is non-inferior to a five day treatment in acute exacerbation of COPD and if total glucocorticoid exposure can be reduced by shorter therapy.

Hypothesis

The investigators postulate, that in an outpatient setting, where generally less severe exacerbations are being treated, a three day treatment duration of systemic corticosteroids should be non-inferior to a five day treatment duration with regard to treatment benefits but decrease cumulative corticosteroid exposure.

Design and Setting

This study is going to be performed as a prospective, randomized, double-blind, placebo-controlled, non-inferiority trial in an outpatient setting. Randomization will be performed as block randomization with a 1:1 allocation. The investigators are going to recruit GPs in northwestern and central Switzerland.

Methods

The investigators are going to include patients presenting to GP's with acute exacerbation of COPD. When matching the investigators eligibility criteria and written informed consent is given, patients included in the study are receiving systemic corticosteroid treatment (equivalent of 40mg prednisone daily) for either five days (conventional arm) or three days (interventional arm) followed by two days of placebo for the interventional group. Pre-randomized, identically looking, numbered blisters are given to all patients included in the study. Antibiotic treatment (Amoxicillin/Clavulanic acid, 625mg 3/d, for ten days) is given to all patients with a CRP ≥50mg/l, COPD and known diagnosis of bronchiectasis, as well as patients presenting with all three of the following symptoms: change of baseline dyspnea, change of sputum quantity and sputum purulence. Further initial treatment and steroid treatment after inclusion is determined and documented by the GP. Patients will undergo follow-up visits at day three and seven by their GP as well as follow-up phone calls executed by the study center at day 30, 90 and 180.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age ≥40 years
* History of ≥10 pack-years of smoking (past or present smokers)
* Airway obstruction, defined as FEV1/FVC≤70%
* Current acute exacerbation of COPD by clinical criteria, defined by the presence of at least two of the following:

  * Change of baseline dyspnea
  * Change of cough
  * Change of sputum quantity or purulence

Exclusion Criteria:

* Diagnosis of asthma
* Initial necessity of hospitalization
* Women who are pregnant or breast feeding
* Premenopausal women with insufficient contraception and anamnestic risk for pregnancy
* Severe coexisting disease with life expectancy <6 months
* Diagnosis of tuberculosis
* Known severe immunosuppression or immunosuppression after solid organ or stem cell transplantation
* Inability to follow study procedures, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study involving an investigational drug
* Previous enrolment into the current study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-03; Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Time to next exacerbation | Six month follow-up period after index exacerbation.

SECONDARY OUTCOMES:
Cumulative glucocorticoid dose | Six month follow-up period after index exacerbation.
Glucocorticoid side effects and complications | Six month follow-up period after index exacerbation.
Change in FEV1 | 7 days follow-up period after index exacerbation.
Hospitalization rate during index exacerbation | Six month follow-up period after index exacerbation.
Overall mortality | Six month follow-up period after index exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg D. Leuppi, Prof., Principal Investigator — Kantonsspital Basleland
Locations (1):
- Kantonsspital Baselland, Liestal, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leuppi JD, Miedinger D, Chhajed PN, Buess C, Schafroth S, Bucher HC, Tamm M. Quality of spirometry in primary care for case finding of airway obstruction in smokers. Respiration. 2010;79(6):469-74. doi: 10.1159/000243162. Epub 2009 Sep 26. PMID 19786731
- [Background] Donaldson GC, Seemungal TA, Bhowmik A, Wedzicha JA. Relationship between exacerbation frequency and lung function decline in chronic obstructive pulmonary disease. Thorax. 2002 Oct;57(10):847-52. doi: 10.1136/thorax.57.10.847. PMID 12324669
- [Background] Makris D, Moschandreas J, Damianaki A, Ntaoukakis E, Siafakas NM, Milic Emili J, Tzanakis N. Exacerbations and lung function decline in COPD: new insights in current and ex-smokers. Respir Med. 2007 Jun;101(6):1305-12. doi: 10.1016/j.rmed.2006.10.012. Epub 2006 Nov 16. PMID 17112715
- [Background] Barnes PJ. Chronic obstructive pulmonary disease. N Engl J Med. 2000 Jul 27;343(4):269-80. doi: 10.1056/NEJM200007273430407. No abstract available. PMID 10911010
- [Background] Sapey E, Stockley RA. COPD exacerbations . 2: aetiology. Thorax. 2006 Mar;61(3):250-8. doi: 10.1136/thx.2005.041822. PMID 16517585
- [Background] Sethi S, Murphy TF. Infection in the pathogenesis and course of chronic obstructive pulmonary disease. N Engl J Med. 2008 Nov 27;359(22):2355-65. doi: 10.1056/NEJMra0800353. No abstract available. PMID 19038881
- [Background] Mohan A, Chandra S, Agarwal D, Guleria R, Broor S, Gaur B, Pandey RM. Prevalence of viral infection detected by PCR and RT-PCR in patients with acute exacerbation of COPD: a systematic review. Respirology. 2010 Apr;15(3):536-42. doi: 10.1111/j.1440-1843.2010.01722.x. PMID 20415983
- [Background] Leuppi JD, Schuetz P, Bingisser R, Bodmer M, Briel M, Drescher T, Duerring U, Henzen C, Leibbrandt Y, Maier S, Miedinger D, Muller B, Scherr A, Schindler C, Stoeckli R, Viatte S, von Garnier C, Tamm M, Rutishauser J. Short-term vs conventional glucocorticoid therapy in acute exacerbations of chronic obstructive pulmonary disease: the REDUCE randomized clinical trial. JAMA. 2013 Jun 5;309(21):2223-31. doi: 10.1001/jama.2013.5023. PMID 23695200
- [Background] Albert RK, Martin TR, Lewis SW. Controlled clinical trial of methylprednisolone in patients with chronic bronchitis and acute respiratory insufficiency. Ann Intern Med. 1980 Jun;92(6):753-8. doi: 10.7326/0003-4819-92-6-753. PMID 6770731
- [Background] Emerman CL, Connors AF, Lukens TW, May ME, Effron D. A randomized controlled trial of methylprednisolone in the emergency treatment of acute exacerbations of COPD. Chest. 1989 Mar;95(3):563-7. doi: 10.1378/chest.95.3.563. PMID 2920584
- [Background] Bullard MJ, Liaw SJ, Tsai YH, Min HP. Early corticosteroid use in acute exacerbations of chronic airflow obstruction. Am J Emerg Med. 1996 Mar;14(2):139-43. doi: 10.1016/S0735-6757(96)90120-5. PMID 8924134
- [Background] Thompson WH, Nielson CP, Carvalho P, Charan NB, Crowley JJ. Controlled trial of oral prednisone in outpatients with acute COPD exacerbation. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):407-12. doi: 10.1164/ajrccm.154.2.8756814.
- [Background] Aaron SD, Vandemheen KL, Hebert P, Dales R, Stiell IG, Ahuja J, Dickinson G, Brison R, Rowe BH, Dreyer J, Yetisir E, Cass D, Wells G. Outpatient oral prednisone after emergency treatment of chronic obstructive pulmonary disease. N Engl J Med. 2003 Jun 26;348(26):2618-25. doi: 10.1056/NEJMoa023161. PMID 12826636
- [Background] Niewoehner DE, Erbland ML, Deupree RH, Collins D, Gross NJ, Light RW, Anderson P, Morgan NA. Effect of systemic glucocorticoids on exacerbations of chronic obstructive pulmonary disease. Department of Veterans Affairs Cooperative Study Group. N Engl J Med. 1999 Jun 24;340(25):1941-7. doi: 10.1056/NEJM199906243402502. PMID 10379017
- [Background] Davies L, Angus RM, Calverley PM. Oral corticosteroids in patients admitted to hospital with exacerbations of chronic obstructive pulmonary disease: a prospective randomised controlled trial. Lancet. 1999 Aug 7;354(9177):456-60. doi: 10.1016/s0140-6736(98)11326-0. PMID 10465169
- [Background] Groenewegen KH, Schols AM, Wouters EF. Mortality and mortality-related factors after hospitalization for acute exacerbation of COPD. Chest. 2003 Aug;124(2):459-67. doi: 10.1378/chest.124.2.459. PMID 12907529
- [Background] Miravitlles M, Mayordomo C, Artes M, Sanchez-Agudo L, Nicolau F, Segu JL. Treatment of chronic obstructive pulmonary disease and its exacerbations in general practice. EOLO Group. Estudio Observacional de la Limitacion Obstructiva al Flujo aEreo. Respir Med. 1999 Mar;93(3):173-9. doi: 10.1016/s0954-6111(99)90004-5. PMID 10464874
- [Background] Walsh LJ, Lewis SA, Wong CA, Cooper S, Oborne J, Cawte SA, Harrison T, Green DJ, Pringle M, Hubbard R, Tattersfield AE. The impact of oral corticosteroid use on bone mineral density and vertebral fracture. Am J Respir Crit Care Med. 2002 Sep 1;166(5):691-5. doi: 10.1164/rccm.2110047. PMID 12204867
- [Background] Decramer M, Lacquet LM, Fagard R, Rogiers P. Corticosteroids contribute to muscle weakness in chronic airflow obstruction. Am J Respir Crit Care Med. 1994 Jul;150(1):11-6. doi: 10.1164/ajrccm.150.1.8025735.
- [Background] Magnussen H, Disse B, Rodriguez-Roisin R, Kirsten A, Watz H, Tetzlaff K, Towse L, Finnigan H, Dahl R, Decramer M, Chanez P, Wouters EF, Calverley PM; WISDOM Investigators. Withdrawal of inhaled glucocorticoids and exacerbations of COPD. N Engl J Med. 2014 Oct 2;371(14):1285-94. doi: 10.1056/NEJMoa1407154. Epub 2014 Sep 8. PMID 25196117
- [Background] Buist AS, McBurnie MA, Vollmer WM, Gillespie S, Burney P, Mannino DM, Menezes AM, Sullivan SD, Lee TA, Weiss KB, Jensen RL, Marks GB, Gulsvik A, Nizankowska-Mogilnicka E; BOLD Collaborative Research Group. International variation in the prevalence of COPD (the BOLD Study): a population-based prevalence study. Lancet. 2007 Sep 1;370(9589):741-50. doi: 10.1016/S0140-6736(07)61377-4. PMID 17765523
- [Background] Jochmann A, Scherr A, Jochmann DC, Miedinger D, Torok SS, Chhajed PN, Tamm M, Leuppi JD. Impact of adherence to the GOLD guidelines on symptom prevalence, lung function decline and exacerbation rate in the Swiss COPD cohort. Swiss Med Wkly. 2012 Apr 5;142:w13567. doi: 10.4414/smw.2012.13567. eCollection 2012. PMID 22481636
- [Background] Anthonisen NR, Manfreda J, Warren CP, Hershfield ES, Harding GK, Nelson NA. Antibiotic therapy in exacerbations of chronic obstructive pulmonary disease. Ann Intern Med. 1987 Feb;106(2):196-204. doi: 10.7326/0003-4819-106-2-196. PMID 3492164
- [Background] Rodriguez-Roisin R. Toward a consensus definition for COPD exacerbations. Chest. 2000 May;117(5 Suppl 2):398S-401S. doi: 10.1378/chest.117.5_suppl_2.398s. PMID 10843984
- [Derived] Urwyler P, Boesing M, Abig K, Cattaneo M, Dieterle T, Zeller A, Bachler H, Markun S, Senn O, Merlo C, Essig S, Ullmer E, Rutishauser J, Schuurmans MM, Leuppi JD. Reduction of corticosteroid use in outpatient treatment of exacerbated COPD - Study protocol for a randomized, double-blind, non-inferiority study, (The RECUT-trial). Trials. 2019 Dec 16;20(1):727. doi: 10.1186/s13063-019-3856-8. PMID 31842993
- See also: 8. The Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2014 — http://www.goldcopd.org